CLINICAL TRIAL: NCT01413906
Title: Phase 1 Multiple Ascending Dose Study of BMS-833923 (XL139) in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA194-010
Record Dates: First submitted 2011-08-04; First posted 2011-08-10 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — BMS-833923

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: BMS-833923 (XL139) (Experimental)
  Interventions: Drug: BMS-833923 (XL139)

INTERVENTIONS:
Drug: BMS-833923 (XL139) — Capsule, Oral, 150 mg, 300 mg, or 450 mg,Once daily, Until progression of disease, unacceptable toxicity, withdrawal of subject's consent or meeting other discontinuation criteria
  Other Names: (XL139)

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety profile of BMS-833923 (XL139) when orally administered on a once daily schedule.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced or metastatic solid tumors refractory to, or relapsed from, standard therapies or for which there is no known effective treatment
* Men and woman, 20 years of age and above

Exclusion Criteria:

* Subjects with symptomatic brain metastasis or active brain metastasis requiring treatments
* Inability to swallow oral medication
* Uncontrolled or significant cardiovascular disease
* Inadequate bone marrow function
* Inadequate hepatic function
* Inadequate renal function
* Pancreatitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLT) and observed adverse events | Within the first 28 days of treatment
Incidence of Dose Limiting Toxicity (DLT) and observed adverse events | Up to 90 days additional treatment period plus 60 days of follow-up

SECONDARY OUTCOMES:
The number of subjects experienced DLT | Within the first 28 days
Maximum observed concentration (Cmax) of BMS-833923 (XL139) | Day1 and Day 29
Trough observed concentration (Cmin) of BMS-833923 (XL139) | Day1 and Day 29
Time of maximum observed concentration (Tmax) of BMS-833923 (XL139) | Day1 and Day 29
Area under the concentration-time curve in one dosing interval [AUC(TAU)] of BMS-833923 (XL139) | Day1 and Day 29
Effective half-life (T-half,eff) of BMS-833923 (XL139) | Day1 and Day 29
Accumulation index (AI) of BMS-833923 (XL139) | Day1 and Day 29
Best overall response assessed according to Response evaluation criteria in solid tumors (RECIST) v1.1 criteria | Up to120 days of treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Kashiwa-shi, Chiba, Japan

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx